CLINICAL TRIAL: NCT04689919
Title: A Single Center, Open Label, Randomized, Single-dose, Two Period Two Way Cross-over Study to Explore the Bioequivalence of Xaroban 20mg (Rivaroxaban) Tablet and Xarelto 20mg (Rivaroxaban) Tablet Under Fed Conditions in Healthy Male Pakistani Subjects.
Brief Title: Bioequivalence of Xaroban 20mg (Rivaroxaban) Tablet and Xarelto 20mg (Rivaroxaban) Tablet Under Fed Conditions
Acronym: Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: The Searle Company Limited Pakistan (Industry); Center for Bioequivalence Studies and Clinical Research (CBSCR), HEJ Research Institute of chemistry, University of Karachi (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-025-RIV-2018/Protocol/1.0
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Two period Two way cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Group [Xarelto 20mg (Rivaroxaban) Tablet] (Active Comparator): Subjects will take their assigned study medication, together with 240 mL of ambient temperature water, at least 1 hour after start of the meal at their scheduled dosing time-point
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet
- Test Group [Xaroban 20mg (Rivaroxaban) Tablet] (Experimental): Subjects will take their assigned study medication, together with 240 mL of ambient temperature water, at least 1 hour after start of the meal at their scheduled dosing time-point
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 20 MG Oral Tablet — The subjects randomly received single oral dose of Rivaroxaban 20 MG Tablet.

SUMMARY:
A single center, open label, randomized, single-dose, two period, Two way cross-over study to explore the Bioequivalence of Test Product Xaroban (Rivaroxaban) 20 mg Tablet with the reference product Xarelto (Rivaroxaban) 20 mg tablet under fed conditions in healthy Pakistani male subjects. Subjects will receive one single dose per treatment period separated by a wash-out period of 7 days. Blood samples will be taken up to 48hours post-dose.

DETAILED DESCRIPTION:
Single oral administrations of study drug in two periods separated by a washout period of 07 days. Subjects will take their assigned study medication orally, together with 240 mL of ambient temperature water, at least 1 hour after start of the meal at their scheduled dosing time-point. Total duration of treatment of study drug will be of 58 hours comprising 10 hours prior drug administration until 48 hours post dose in each study period.

Pharmacokinetic parameters include Rivaroxaban plasma concentrations at the given sampling times. In each period 16 blood samples for plasma Rivaroxaban concentrations will be taken on Day 2, Day 3 and Day 4 including 0.00 hour pre dose and post dose at 0.25, 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 3.5, 4.00, 6.00, 8.00, 12.00, 24.00, 36.00 and 48.00 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years inclusive.
* Subjects with a body mass index from 18.5 to 30 kg/m2 (both inclusive).
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (i.e., blood pressure, heart rate, and temperature), 12 Lead ECG, and laboratory analysis (i.e., hematology, blood biochemistry, and urinalysis), as determined by the investigator.
* Subjects should have negative urine test for drugs of abuse (Opiates, benzodiazepines, amphetamines, barbiturates, cannabinoids and cocaine will be tested) and alcohol breath analysis at screening and prior to each check-in.
* Subjects and their partners are willing to use reliable non-hormonal contraceptive methods (condoms, diaphragm, non-hormonal intra-uterine device (IUD), female or male sterilization or sexual abstinence) throughout the study and up to 30 days after the last administration of the study drug.
* All subjects should be free from any epidemic or contagious diseases (e.g. Malaria, Dengue, Covid-19).
* Subjects will be able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.

Exclusion Criteria:

* History of smoking (≤3cigarette/day), alcoholism, and test for drug of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.
* Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, gastrointestinal (GI) bleeding within 6 months of randomization, history of intracranial, intraocular, spinal or atraumatic intra-articular bleeding, chronic hemorrhagic disorder, known intracranial neoplasm, arteriovenous malformation, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Subjects receiving concomitant systemic treatment with azole-antimycotics (such as ketoconazole, itraconazole, voriconazole and posaconazole) or HIV protease inhibitors (e.g., ritonavir).
* Subjects receiving NSAIDs (including acetylsalicylic acid) and platelet aggregation inhibitors as these medicinal products typically increase the bleeding risk.
* Subjects receiving concomitant P-gp inhibitor (Erythromycin, Clarithromycin and Azithromycin).
* The concomitant use of rivaroxaban with other strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, phenobarbital or St. John's Wort (Hypericum perforatum).
* Subject with known coagulation disorders (e.g. von Willebrand's disease, hemophilia)
* Subject with known disorders with increased bleeding risk (e.g. periodontosis, hemorrhoids, acute gastritis, peptic ulcer).
* Subject with known sensitivity to common causes of bleeding (e.g. nasal).
* Individuals with mild (creatinine clearance 50 - 80 ml/min), moderate (creatinine clearance 30 - 49 ml/min) and severe (creatinine clearance 15 - 29 ml/min) renal impairment.
* Subject is allergic to Rivaroxaban and/or other Factor Xa inhibitors.
* Subject has received any investigational drug within four weeks.
* Subjects with significant hepatic disease (including moderate to severe hepatic impairment, i.e. Child-Pugh B and C) which is associated with coagulopathy leading to a clinically relevant bleeding risk.
* Subjects with cardiac related conditions (hemodynamically significant mitral valve stenosis, prosthetic heart valve, planned cardioversion, transient atrial fibrillation caused by reversible disease Subjects with known presence of atrial myxoma or left ventricular thrombus and active endocarditis.[8]
* Subjects with salt imbalance in the blood (especially low levels of potassium or magnesium in the blood)
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* Ingestion of OTC drug, within 7 days of drug administration.
* History of intake of any prescribed medicine during a period of 30 days, prior to drug administration day of study.
* History of any significant illness in the last four weeks
* Consumption of grapefruit and/or its products within 14 days prior to the start of study.
* Vitamin, dietary supplements and herbal products must be discontinued 14 days prior to the first dose of study medication.
* Subjects who test positive for syphilis (VDRL) or who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2).
* Individuals having undergone any major surgery within 3 months prior to the start of the study, unless deemed eligible, otherwise by the Principal Investigator or whomever he/she may designate.
* Subject has a history of any illness that, in the opinion of investigator might confound the result of the study or post additional risk in administrating Rivaroxaban to the subject.
* Inability to take oral medication.
* Subjects with any condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or elimination of drugs.
* Subjects testing positive for COVID-19 or are known to have such family members who tested positive for COVID-19 in recent times will also be excluded.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-19 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 2 weeks
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 2 weeks
  plasma concentration-time curve from zero to the time of the last measurable time point t
Area under the plasma concentration versus time curve (AUC)0-∞ | 2 weeks
  area under the plasma concentration-time curve from zero to infinity

OTHER OUTCOMES:
maximum plasma concentration (tmax) | 2 weeks
  time to reach the maximum plasma concentration after drug administration (tmax)
Incidence of Treatment-Emergent Adverse Events | During 2 weeks
  Collection of adverse events
Incidence of abnormal blood pressure | 2 weeks
  Monitor the blood pressure
Incidence of abnormal temperature | 2 weeks
  Monitor the temperature
Incidence of abnormal pulse | 2 weeks
  Monitor the pulse
Incidence of abnormal electrocardiogram waveform | 2 weeks
  Electrocardiogram inspection for QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Raza Shah, PhD, Principal Investigator — CBSCR , ICCBS, University of Karachi; Naghma Hashmi (Co-PI), PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR), ICCBS, university of Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by The Searle Co., Ltd. and the research center (CBSCR).
  The information can not be disclosed or distributed in any way without the written permission of the General Manager of CBSCR-ICCBS & The Searle Company.